CLINICAL TRIAL: NCT02263300
Title: Does Spatial Orientation Affect the Rate of Learning Fiberoptic Intubation Skills in the Novice: A Randomized Controlled Trial
Brief Title: Spatial Orientation and Fiberoptic Intubation Skills in the Novice: A Randomized Controlled Trial
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Raymond Glassenberg, Principal Investigator, Northwestern University
Other Study IDs: STU00098465
Record Dates: First submitted 2014-09-24; First posted 2014-10-13 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Airway Management
Keywords: Fiberoptic Intubation; Medical student; Virtual larynx; Didactic Training; Medical Education

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Supine- Supine: Group A (supine-supine) will first practice fiberoptic intubation with the iLarynx oriented in the supine position. Learning curves, global rating scale and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the SUPINE then UPRIGHT position. At the end of one week,the same medical student will then perform the intubation with the mannequin in both positions.
- Upright-upright: Group B (upright-upright) will first practice fiberoptic intubation with the iLarynx oriented in the upright position. Learning curves, global assessment score and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the UPRIGHT then SUPINE position.At the end of one week, the same medical student will then perform the intubation with the mannequin in both positions.
- Supine -upright: Group C( supine -upright) will first practice fiberoptic intubation with the iLarynx oriented in the supine position. Learning curves, global assessment score and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the UPRIGHT then SUPINE position. At the end of one week, The same medical student will then perform the intubation with the mannequin in both positions.
- Upright - supine: Group D( upright - supine) will first practice fiberoptic intubation with the iLarynx oriented in the upright position. Learning curves, global assessment score and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the SUPINE then UPRIGHT position. At the end of one week, the same medical student will then perform the intubation with the mannequin in both positions.

SUMMARY:
Does spatial orientation of a novice in relation to a mannequin (supine vs upright) impact on the development of fiberoptic intubation skills?

Is it necessary to teach both orientations or is the supine view transferable to the upright position?

Which method demonstrates longer skill retention?

The hypotheses: Both orientations must be practiced and the upright skill is harder to learn but is retained for longer.

DETAILED DESCRIPTION:
Following IRB approval, written consent to participate in the study will be obtained from medical students

Phase one :

Forty medical students, novices in fiberoptic intubation use will be recruited and randomly assigned into one of two groups:

Group A (supine-supine) will first practice fiberoptic intubation with the iLarynx oriented in the supine position. Learning curves, global rating scale and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the SUPINE then UPRIGHT position. At the end of one week,the same medical student will then perform the intubation with the mannequin in both positions.

Group B (upright-upright) will first practice fiberoptic intubation with the iLarynx oriented in the upright position. Learning curves, global assessment score and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the UPRIGHT then SUPINEposition.At the end of one week, the same medical student will then perform the intubation with the mannequin in both positions.

Group C( supine -upright) will first practice fiberoptic intubation with the iLarynx oriented in the supine position. Learning curves, global assessment score and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the UPRIGHT then SUPINE position. At the end of one week, The same medical student will then perform the intubation with the mannequin in both positions.

Group D( upright - supine) will first practice fiberoptic intubation with the iLarynx oriented in the upright position. Learning curves, global assessment score and checklist will then be obtained by a blinded examiner with the medical student using a real fiberoptic on a mannequin oriented in the SUPINE then UPRIGHT position. At the end of one week, the same medical student will then perform the intubation with the mannequin in both positions.

teaching testing testing week testing testing

Group A supine supine upright random random random random B upright upright supine random random random random C supine upright supine random random random random D upright supine upright random random

Phase two:

Study candidates will randomly be assigned(20 per group) to practice for 15minutes/day their intubations skills with the iLarynx application downloaded to their smart phones or iPads. The other group (20candidates) will be asked not to practice their intubation skills. At the end of one week both groups will be retested on a mannequin by the same blinded examiner to obtain a new learning curve, global assessment score and checklist. Both orientations of the mannequin will be tested and the order randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* Third and fourth year medical student
* no previous training in fiberoptic intubation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Third and fourth year medical students.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03-30 (Actual); Study Completion 2015-03-30 (Actual)

PRIMARY OUTCOMES:
Elapsed time to mannequin intubation with fiberoptic scope. | 2 minutes
  The elapsed time of intubation with fiberoptic scope of a mannequin. Stop watch is started at passing teeth and ends when scope reaches carina.

SECONDARY OUTCOMES:
Global rating scale (GRS) | 2 minutes
  Global rating scale (GRS) and assessment of medical students skill demonstrated during fiberoptic intubation of a mannequin on a score of 1-5 1 being very poor and 5 being clearly superior.
Examiner check list (ECL) scores | 2 mintues
  The ECL will be used to measure the students proficiency with the fiberoptic scope on a scale of 0-5 for each attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Glassenberg, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badurdeen S, Abdul-Samad O, Story G, Wilson C, Down S, Harris A. Nintendo Wii video-gaming ability predicts laparoscopic skill. Surg Endosc. 2010 Aug;24(8):1824-8. doi: 10.1007/s00464-009-0862-z. Epub 2010 Jan 28. PMID 20108147
- [Background] Boet S, Bould MD, Schaeffer R, Fischhof S, Stojeba N, Naik VN, Diemunsch P. Learning fibreoptic intubation with a virtual computer program transfers to 'hands on' improvement. Eur J Anaesthesiol. 2010 Jan;27(1):31-5. doi: 10.1097/EJA.0b013e3283312725. PMID 19851113
- [Background] De Oliveira GS Jr, Glassenberg R, Chang R, Fitzgerald P, McCarthy RJ. Virtual airway simulation to improve dexterity among novices performing fibreoptic intubation. Anaesthesia. 2013 Oct;68(10):1053-8. doi: 10.1111/anae.12379. Epub 2013 Aug 19. PMID 23952805
- [Background] Goldmann K, Steinfeldt T. Acquisition of basic fiberoptic intubation skills with a virtual reality airway simulator. J Clin Anesth. 2006 May;18(3):173-8. doi: 10.1016/j.jclinane.2005.08.021. PMID 16731318
- [Background] Chandra DB, Savoldelli GL, Joo HS, Weiss ID, Naik VN. Fiberoptic oral intubation: the effect of model fidelity on training for transfer to patient care. Anesthesiology. 2008 Dec;109(6):1007-13. doi: 10.1097/ALN.0b013e31818d6c3c. PMID 19034097
- [Background] Marsland CP, Robinson BJ, Chitty CH, Guy BJ. Acquisition and maintenance of endoscopic skills: developing an endoscopic dexterity training system for anesthesiologists. J Clin Anesth. 2002 Dec;14(8):615-9. doi: 10.1016/s0952-8180(02)00456-7. PMID 12565124

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT02263300/Prot_SAP_000.pdf